CLINICAL TRIAL: NCT04255069
Title: A Phase 2, Randomized, Multiple-Dose, Double-Blind, Placebo-Controlled Study of JKB-122 in Patients With Non-Alcoholic Steatohepatitis (NASH) and Fibrosis
Brief Title: A Study to Evaluate the Efficacy and Safety of JKB-122 in Patients With NASH and Fibrosis
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: TaiwanJ Pharmaceuticals Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: TWJ-NAF
Record Dates: First submitted 2020-01-24; First posted 2020-02-05 (Actual); Last update posted 2020-02-13 (Actual); Status verified 2020-02

CONDITIONS: Nonalcoholic Steatohepatitis (NASH) With Fibrosis
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease | interventions — JKB-122

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Placebo (Placebo Comparator): Placebo, oral, daily
  Interventions: Drug: Placebo
- Dose 1 (Experimental): JKB-122, Dose 1, oral, daily
  Interventions: Drug: Dose 1 JKB-122
- Dose 2 (Experimental): JKB-122, Dose 2, oral, daily
  Interventions: Drug: Dose 2 JKB-122

INTERVENTIONS:
Drug: Placebo — A treatment with dose 1 JKB-122, dose 2 JKB-122 or placebo will be randomly administrated once daily
  Arms: Placebo
Drug: Dose 1 JKB-122 — A treatment with dose 1 JKB-122, dose 2 JKB-122 or placebo will be randomly administrated once daily
  Other Names: JKB-122
  Arms: Dose 1
Drug: Dose 2 JKB-122 — A treatment with dose 1 JKB-122, dose 2 JKB-122 or placebo will be randomly administrated once daily
  Other Names: JKB-122
  Arms: Dose 2

SUMMARY:
A double-blind placebo controlled randomized Phase 2 study to determine if JKB-122 compared with placebo resolves NASH on liver biopsy and improves fibrosis

DETAILED DESCRIPTION:
This is a Phase 2 study in which JKB-122 is given once daily for 52 weeks to subjects with Nonalcoholic steatohepatitis (NASH) with Fibrosis who have biopsy reading more than NAS 4 with a fibrosis reading more than 1 and no cirrhosis. Subjects will be at least 18 years of age, either male or female.

ELIGIBILITY:
Inclusion Criteria:

1. Is male or female, 18 years to 70 years of age.
2. If female of childbearing potential, must not be pregnant or breastfeeding and either postmenopausal (no menses for previous 12 months) or using an effective method of birth control (e.g., oral contraceptives, hormonal injectable or implanted contraceptives, tubal ligation, or partner with vasectomy plus a barrier method).
3. Is diagnosed with non-alcoholic steatohepatitis (NASH) NAS >4.0
4. Compensated liver disease with the following hematologic, biochemical, and serological criteria on entry into protocol:
5. Subjects taking lipid lowering agents should keep their dose stable during the study.
6. Stable use of insulin sensitizing agents (PPARs, SGLT2 inhibitors, or GLP-1 agonists for 6 months prior to screening liver biopsy).
7. Is capable of understanding and signing the informed consent document. If subject is unable to sign the informed consent form, then the subject's legal representative or guardian may provide written consent per local regulations.
8. Agrees to comply with protocol requirements.

Exclusion Criteria:

1. Has human immunodeficiency virus (HIV) or is hepatitis B or C positive.
2. Has history of liver cirrhosis.
3. Has glycated hemoglobin (HbA1c ) greater than 9%.
4. Binge drinking as drinking 5 or more alcoholic drinks
5. Significant alcohol consumption
6. Is being treated with any prescription narcotic drug (including transdermal delivery systems).
7. Has a known or suspected central nervous system disorder that may predispose to seizures or lower the seizure threshold.
8. Has unstable and uncontrollable hypertension (>180/110 mmHg).
9. Has received other therapies for NAFLD in the last 4 weeks prior to the screening visit (Day -7).
10. Requires concomitant use of or treatment with opioids or other excluded drugs such as hepatotoxic medications.
11. Has received other investigational agents within 30 days prior to the screening visit (Day -7).
12. Has either autoimmune or genetic liver disease.
13. Alpha- fetoprotein greater than 20 mcg/L. Has impaired renal function (i.e. serum creatinine CLcr < 60 mL/min).
14. Subjects who gained or lost weight greater than 5 kg in the past 3 months.
15. Any form of chronic liver disease other than NASH
16. Suspected or confirmed cirrhosis. -

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2020-06-30 (Estimated); Primary Completion 2023-06-30 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
To evaluate the effect of JKB-122 compared to placebo to achieve NASH resolution on liver histology in non-cirrhotic NASH patients with stage 2 or 3 fibrosis | 52 weeks
  Assessment will be based on the proportion of JKB-122 15 mg or 35 mg treated patients relative to placebo achieving NASH resolution with at least a 2 point reduction in NAS and no worsening of fibrosis
To evaluate the effect of JKB-122 compared to placebo to achieve a ≥ 1 stage fibrosis improvement on liver histology in non-cirrhotic NASH patients with stage 2 or 3 fibrosis | 52 weeks
  Assessment will be based on the proportion of JKB-122 15 mg or 35 mg treated patients relative to placebo achieving at least a 1 stage improvement in fibrosis (NASH Clinical Research Network system) by liver biopsy with no worsening of NAS.

SECONDARY OUTCOMES:
Evaluate the changes of hepatic fat content | 52 weeks
  The changes of fatty liver content (%) will be measured by MRI-PDFF.
Evaluate the changes of fibrosis score | 52 weeks
  The changes of fibrosis score (kPa) will be measured by FibroScan.

IPD SHARING:
Plan to Share IPD: No